CLINICAL TRIAL: NCT02754778
Title: Evaluation of Practicability in Survey and Test Procedures and of Successful Implementation of Complex Interventions - Feasibility Analysis Based on a Pilot Study: Influence of Conditional Workout Postpartum on Arterial Stiffness Among Women With Status After Preeclampsia, Superimposed Preeclampsia or HELLP-syndrome
Brief Title: Influence of Conditional Workout Postpartum on Arterial Stiffness Among Women With Status After Preeclampsia, Superimposed Preeclampsia or HELLP-syndrome
Acronym: RedCarRisk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Gregor Seliger, Dr. med. Gregor Seliger, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RedCarRisk-Study
Record Dates: First submitted 2016-04-22; First posted 2016-04-28 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Preeclampsia; Superimposed Preeclampsia; HELLP Syndrome
Keywords: arterial stiffness; preeclampsia; HELLP-syndrome; pulse wave velocity; advanced glycation endproducts; skin autofluorescence; conditional workout; postpartum; cardiovascular risk; pregnancy; vicorder; age reader
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): no intervention, regular family life
- intervention group (Active Comparator): 6 month of regular conditional workout 1-3 times a week
  Interventions: Behavioral: conditional workout

INTERVENTIONS:
Behavioral: conditional workout — 6 month of regular conditional workout 1-3 times a weak
  Arms: intervention group

SUMMARY:
Evaluation of practicability in survey and test procedures and of successful implementation of complex interventions - feasibility analysis based on a pilot study: Influence of conditional workout postpartum on arterial stiffness among women with status after preeclampsia, superimposed preeclampsia or HELLP-syndrome

DETAILED DESCRIPTION:
Cardiovascular disease is the main cause of death among women in Europe and in the USA. Its costs amount annually more than 196 billions Euro in Europe. The federal state of Saxony-Anhalt occupies leading position in mortality in myocardial infarction and coronary heart disease in Germany. Up to 8 percent of all pregnant women develop a severe pregnancy-associated hypertension, like preeclampsia, superimposed preeclampsia or HELLP-syndrome. These women have an increased lifetime risk for cardio- and cerebrovascular diseases.

The consecutive increasing arterial stiffness because of endothelial dysfunction is a determining factor in etiology of pregnancy-associated hypertension and results in increased cardiovascular risk. Aortal pulse wave velocity is used as Goldstandard for measuring arterial stiffness.

Pregnant women suffering from a severe pregnancy-associated hypertension present higher levels in arterial stiffness measured by pulse wave velocity than healthy pregnant women. Pathological changes of the vascular systems persistent from 6 month until 10 years after delivery and give an explanatory approach for an increased cardiovascular longterm risk at these patients. Numerous medical associations like American Heart Association aim at reducing especially cardiovascular longterm risk in women with status after preeclampsia, superimposed preeclampsia or HELLP syndrome.

Pregnancy-independent studies in patients with coronary heart disease and analysis in women with metabolic syndrome show a reduction of arterial stiffness by regular conditional workout.

Scientific problem of this pilot study: If a reduction in arterial stiffness in women from a risk group - during a 6-month-ongoing intensive regular conditional workout within a midwife-supported teamwork and under inclusion of dietary interventions - achieved?

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of preeclampsia, superimposed gestosis or HELLP syndrome
* capacity for content

Exclusion Criteria:

* eclamptic stroke
* New York Heart Association > Stadium II
* severe neurological or orthopedic disabilities
* peripheral arterial occlusive disease
* severe disease of the newborn which leads to an intensive familial care

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
reduced aortic pulse wave velocity by 1m/s | six month

SECONDARY OUTCOMES:
no arterial hypertension defined as blood pressure ≤140mmHg / 80mmHg without antihypertensic medication | 13 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Riemer, Dr. med., Principal Investigator — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg; Gregor Seliger, Dr. med., Principal Investigator — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg
Locations (2):
- Germany (2):
  - St. Elisabeth and St. Barbara Hospital / Women's clinic, Halle, Saint
  - Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Paper — https://www.thieme-connect.com/products/ejournals/html/10.1055/a-1345-8733?articleLanguage=en